CLINICAL TRIAL: NCT05614427
Title: The LAVA (Lateral Flow Antigen Validation and Applicability) 2 Study for COVID-19
Acronym: LAVA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 292509
Record Dates: First submitted 2022-11-09; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior nasal swab (Active Comparator): Lateral flow tests performed on anterior nasal swabs compared to routinely taken nose and throat swabs with RT-PCR
  Interventions: Diagnostic Test: Innova Lateral Flow Test
- Buccal swab (Active Comparator): Lateral flow tests performed on buccal swabs compared to routinely taken nose and throat swabs with RT-PCR
  Interventions: Diagnostic Test: Innova Lateral Flow Test

INTERVENTIONS:
Diagnostic Test: Innova Lateral Flow Test — Lateral flow test performed on anterior nasal or buccal swabs

SUMMARY:
The Lateral Flow Antigen Validity and Applicability (LAVA) 2 study aims to determine the validity of lateral flow antigen devices (LFDs) used to perform point of care testing for COVID-19, compared to the current gold standard test of RTPCR in children. In a pilot study we have shown that the anterior nose swabs used to perform a LFD test are associated with significantly lower pain scores than the nose and throat swabs used to perform RT-PCR tests and that the results are available significantly more quickly. RT-PCR is an excellent diagnostic test but one drawback includes remaining positive for a prolonged period, potentially when the person is no longer infective, as it can pick up viral particulate rather than live virus. LFDs are more likely to be positive at the point that a person has a high viral load and is therefore infectious to others, but this has not been studied in non-laboratory settings in children. The study aims to determine the correlation between LFD and viral load detected on RT-PCR in children to enable the utility of the test in different clinical and non-clinical settings to be better determined.

DETAILED DESCRIPTION:
Purpose and Design This study aims to answer key questions about testing for COVID-19 in children. COVID-19 in children is very different from adults: COVID-19 infection is less prevalent in children compared to adults and the disease course is very much milder, with children being more likely to be asymptomatic than adults. Currently, all children admitted to hospital or undergoing a procedure under general anaesthetic are routinely tested for SARS-CoV-2 using RT-PCR performed on a nose and throat swab. Whilst this is an excellent diagnostic test for someone who is symptomatic with COVID-19, it can remain positive for a significant period after a person has been infected with COVID-19 and is no longer a risk to others. In a clinical setting this can result in elective operations being cancelled, potentially unnecessarily. Additionally, it means that children who may be infective with COVID-19 are less likely to be symptomatic with the infection, indeed many patients who have been diagnosed with COVID-19 have been admitted to hospital for an unrelated cause, making differentiation on the basis of symptoms difficult. We have chosen to look primarily at the relationship between lateral flow device tests performed on anterior nasal swabs, which are a less painful swab and give a rapid result, compared to the viral load detected using RT-PCR performed on a nose and throat swab. This will complement ongoing work which is being performed outside of the group proposing this study, which is examining the relationship between viral load and infectivity. This study will be able to determine the performance of the LFD at different viral loads and therefore the utility of the LFD within clinical settings to predict which patients are infective with SARS-CoV-2.

The study has been designed by a multidisciplinary team, described in the steering group. Unfortunately due to the need to deliver this study rapidly, patient and parental input has not been specifically sought but the pain scores described in the pilot study work display the acceptability of this test to parents.

Recruitment and consent In order to recruit a sufficient number of patients to answer the study question in a timely way, as is required, we have built into the protocol the option to take deferred consent to participate in the study. The acceptability of the swabs is clear within the pilot study and the test is being widely used in community settings already. Deferred consent is not felt to be appropriate for children in the peri-operative period due to the impact that it may have on their clinical care and therefore patients and families will be approached about the study before the swab is performed. In all other settings, a routine swab for SARS-CoV-2 is being performed anyway which is more painful for the child than the study swab.

The specificity of the LFD has been shown to be very good (99.6%) in laboratory and clinical settings and therefore employing the use of the LFD within the study may also enable hospitals to detect asymptomatic infective children with COVID-19 earlier in their admission. A recording of the patients who are approached before a routine swab is performed but who decline the test will be kept to ensure that a swab is not performed anyway with the assumption that they will be approached for deferred consent. The record will include the child's hospital number and the parent's email address. No additional details will be held. Patients will be approached for consent by being emailed a small amount of information about the study with a link to the PIS followed by a link to the consent form, with the option to record refusal of consent if they do not wish to participate. The appropriate PISC will be sent according to whether they are approached before or after the anterior nose swab has been taken. The person emailing the patients the PISC does not have to be GMP trained, but should a patient or their family wish to ask questions they will have the details of the study team's telephone number and email address. Inclusion/exclusion This study is intended to include all children under 18 years of age who are undergoing routine swabbing or who are having a procedure performed under general anaesthetic. Risks, burdens and benefits Having undertaken the pilot study we have had opportunity to understand the impact on patients and their families.

Many patients and parents were positive about participating in the study, appreciating the opportunity to have an additional test prior to an operation and getting the results of the LFD test back more quickly. As shown in the pilot study, the pain scores given by children and parents were significantly lower using anterior nasal swabs compared to nose and throat swabs suggesting that there is much higher acceptability of the test. Some participants did refuse to participate because they were concerned that their child may find an additional swab distressing or because they did not want to run the risk of a long-awaited elective procedure being cancelled. During the pilot study we found no adverse events associated with the anterior nasal swabs and given the lower pain scores seen, can reassure parents that the swab required for the LFD is significantly less painful for a child. Confidentiality We are collecting the hospital number of each patient to enable accurate tracking of patients within the study. These will be visible to the central study team but each site's patients will only be visible to patients within that site. The first half of the postcode is being collected because subsequent analysis of the positive predictive value of the test requires the prevalence of COVID-19 to be known. The DOB and sex of the child is being collected so that the demographics of the patients included in the study are known, enabling appropriate conclusions to be drawn. CAG approval has not been sought as the COPI notice issued by the Secretary of State allows the appropriate collection of data within studies focussed on COVID-19 to be collected and can include people who do not sit within the direct care team to contribute to the recruitment and running of the study. Conflict of interest None of the study group have any declared conflict of interest in the study. The results will be given to Public Health England and will be submitted for peer review and subsequent publication.

ELIGIBILITY:
Inclusion Criteria:

* Child undergoing routine RT-PCR testing for SARS-CoV-2 using a nose and throat or ET sample
* Child with positive RT-PCR for SARS-CoV-2 within the last 72 hours

Exclusion Criteria:

* None

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
The association of LFD result (positive/negative) taken from an anterior nares swab compared to RT-qPCR finding (Cycle Threshold Values) | Swabs will be taken within 30 minutes of each other
The association of LFD result (positive/negative) taken from a buccal swab compared to RT-qPCR finding (Cycle Threshold Values) | Swabs will be taken within 30 minutes of each other

SECONDARY OUTCOMES:
The overall sensitivity of the LFD compared to RT-PCR. | Swabs will be taken within 30 minutes of each other
The overall specificity of the LFD compared to RT-PCR. | Swabs will be taken within 30 minutes of each other

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No